CLINICAL TRIAL: NCT00426439
Title: Chloroquine and Coartem for Treatment of Symptomatic Children With Plasmodium Falciparum in Guinea Bissau.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Responsible Party: Dr. Poul-Erik Kofoed, Bandim Heath Project
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSB-2006-Coartem
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Malaria, Falciparum
Keywords: malaria; Plasmodium falciparum; children; Guinea-Bissau; artemether; lumefantrine; chloroquine; Coartem
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Chloroquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Coartem (Experimental): Treatment of documented malaria in children following the dosages recommended by the manufacturer.
  Interventions: Drug: Chloroquine; Drug: Artemether-lumefantrine (Coartem)
- 2 Chloroquine (Active Comparator): The antimalarial actually used in Guinea-Bissau is the dosage of 50 mg/kg given twice a day for 3 days.
  Interventions: Drug: Chloroquine; Drug: Artemether-lumefantrine (Coartem)

INTERVENTIONS:
Drug: Chloroquine — Chloroquine tablets gives as 50 mg/kg divided into 6 doses giver twice a day for 3 days.
Drug: Artemether-lumefantrine (Coartem) — Will be dosed according to the recommendations of WHO. Will be given at time: 0 h, 8 h, 24 h, 36 h,48 h and 60 h. The dosage will be according to bodyweight of the child as follows: 5-14 kg: 1 tablet, 15-24 kg: 2 tablets, 25-34 kg: 3 tablets, < 34 kg: 4 tablets.
  Other Names: Brand name: Coartem.

SUMMARY:
This study will evaluate the efficacy of treatment with artemether-lumefantrine as compared to chloroquine in the dose of 50 mg/kg for treatment of malaria in children in Guinea-Bissau. The genetic basis of the parasites for developing resistance will be examined. Children coming to one of the Health Centres with symptoms of malaria and a positive malaria test will be included. The children will be followed weekly until day 70. In case of reappearance of parasites the child will be re-treated with the opposite study drug.

DETAILED DESCRIPTION:
This study compares treatment of uncomplicated malaria in children in Guinea-Bissau with artemether-lumefantrine (Coartem) with that of treatment with chloroquine 50 mg/kg. Furthermore, the genetic basis of anti-malarial resistance in Guinea-Bissau will be studied by analyzing specific single nucleotide polymorphisms in pfcrt and pfmdr1 in blood samples from this in vivo trial. We also intend to study whether the recent report that chloroquine sensitive parasites are selected at recrudescence after Coartem is confirmed in Bissau.

Following consent to participate, children visiting one of the Health Centres in the study area with mono-infection with Plasmodium falciparum are by block-randomization allocated to one of the treatment groups. The treatment is given supervised by one of the health workers and malaria film taken on day 2 and 3. The children are visited and malaria films obtained once weekly until day 70. On day seven, 100 microliter of capillary blood are drawn for analyses of analyses of drug concentrations in whole blood. On inclusion and whenever a child has recurrent parasitaemia, a filter-paper blood-sample is collected for later PCR analysis. On the day of inclusion, on day 42 and on day 70 the haemoglobin level is measured.

If parasites reappear in 50% or more of at least 40 children in one of the treatment groups this treatment arm should be terminated. During the study parents are recommended to bring the child to the health centre in case of any illness. Participating children will be examined and treated free of charge. The opposite study drug will be used for re-treatment of children in case of recrudescence, and the child will be followed as previously planned.

The results from this study could be used for the planning of the recommendations for treatment of malaria in Guinea-Bissau. It will provide the National Malaria Programme with information of the efficacy of Coartem before it is implemented.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting at one of the health centres in the study area
* Symptoms suggestive of malaria
* At least 20 P.falciparum parasites per 200 leucocytes
* Living in the study area (to enable follow-up)

Exclusion Criteria:

* Danger signs
* By the responsible doctor evaluated to need to be transferred to the national hospital as an in-patient
* Previous idiosyncratic reactions to any of the study drugs

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Parasite reappearance rate, | 70 days

SECONDARY OUTCOMES:
genetic markers of resistance | 70 days
recrudescence and re-infection rates | 70 days
Hospitalisation during follow-up | 70 days
Haemoglobin changes | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau Region, Guinea-Bissau

REFERENCES:
- [Derived] Jovel IT, Kofoed PE, Rombo L, Rodrigues A, Ursing J. Temporal and seasonal changes of genetic polymorphisms associated with altered drug susceptibility to chloroquine, lumefantrine, and quinine in Guinea-Bissau between 2003 and 2012. Antimicrob Agents Chemother. 2015 Feb;59(2):872-9. doi: 10.1128/AAC.03554-14. Epub 2014 Nov 24. PMID 25421474
- [Derived] Ursing J, Kofoed PE, Rodrigues A, Blessborn D, Thoft-Nielsen R, Bjorkman A, Rombo L. Similar efficacy and tolerability of double-dose chloroquine and artemether-lumefantrine for treatment of Plasmodium falciparum infection in Guinea-Bissau: a randomized trial. J Infect Dis. 2011 Jan 1;203(1):109-16. doi: 10.1093/infdis/jiq001. PMID 21148503